CLINICAL TRIAL: NCT05061771
Title: A Randomized, Part A Partial Blinded and Part B Double Blinded, Placebo-controlled 24-week Clinical Study to Evaluate the Efficacy and Safety of Nomacopan Therapy in Adult Patients With Bullous Pemphigoid Receiving Adjunct Oral Corticosteroid Therapy (ARREST-BP)
Brief Title: Nomacopan Therapy in Adult Patients With Bullous Pemphigoid Receiving Adjunct Oral Corticosteroid Therapy (ARREST-BP)
Acronym: ARREST-BP
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Akari has decided to discontinue AK802 study due to strategic resource allocation decisions.
Sponsor: AKARI Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK802
Record Dates: First submitted 2021-09-15; First posted 2021-09-30 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2022-10

CONDITIONS: Bullous Pemphigoid
Keywords: pemphigoid; blistering skin disease; nomacopan; complement; leukotriene
MeSH Terms: conditions — Pemphigoid, Bullous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- nomacopan (rVA576) (Active Comparator): PART A:
  High dose nomacopan (standard complement ablating doses on Day 1 followed by 45 mg qd) administered by subcutaneous injection, plus a starting dose of 0.5 mg/kg/day OCS qd
  or
  Low dose nomacopan (standard complement ablating doses on Day 1 followed by 15 mg qd) administered by subcutaneous injection, plus a starting dose of 0.5 mg/kg/day OCS
  PART B:
  Nomacopan (standard complement ablating doses on Day 1 followed by to be confirmed mg qd) administered by subcutaneous injection, plus a starting dose of 0.5 mg/kg/day OCS qd
  Interventions: Drug: nomacopan (rVA576)
- Placebo (Placebo Comparator): PART A:
  Placebo (matching standard complement ablating doses on Day 1 and then matching injection volume of 45mg dose qd) administered by subcutaneous injection, plus a starting dose of 0.5 mg/kg/day oral corticosteroid (OCS) qd
  or
  Placebo (matching standard complement ablating doses on Day 1 and then matching injection volume of 15mg dose qd) administered by subcutaneous injection, plus a starting dose of 0.5 mg/kg/day oral corticosteroid (OCS) qd
  PART B:
  Placebo (matching standard complement ablating doses on Day 1 and then matching injection volume of active dose qd) administered by subcutaneous injection, plus a starting dose of 0.5 mg/kg/day oral corticosteroid (OCS) qd
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: nomacopan (rVA576) — Nomacopan an inhibitor of complement C5 and LTB4
  Arms: nomacopan (rVA576)
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
A phase III two-part study of nomacopan, a bifunctional inhibitor of complement component C5 and leukotriene B4 (LTB4), for the treatment of moderate and severe bullous pemphigoid. There is evidence that both terminal complement activation (via C5) and the lipid mediator LTB4 may have a central role in driving the disease. In this study patients will be randomized to receive either nomacopan plus oral corticosteroids (OCS) or placebo plus OCS for a treatment period of 24 weeks. OCS will be tapered over the course of the treatment if the symptoms of disease improve.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between 18 and 89 years of age inclusive at the time of consent with Karnofsky score of 50% or more at screening
2. Male or female ≥90 years of age at the time of consent with Karnofsky score of 70% or more at screening
3. Diagnosis of Bullous Pemphigoid either newly diagnosed or relapsing
4. Patients with confirmed atypical Bullous Pemphigoid
5. Bullous Pemphigoid classified as either moderate or severe on the basis of the Investigator Global Assessment (IGA) at randomisation
6. Willing to receive immunisation against Neisseria meningitidis and/or antibiotic prophylaxis
7. Provision of voluntary written informed consent

Exclusion Criteria:

1. Patients with recalcitrant BP that have never achieved CDA or who have never been in complete disease remission despite long term treatment with super potent topical steroid or oral cotricosteroid
2. Epidermolysis bullosa acquisita, mucous membrane pemphigoid, or anti p200 pemphigoid
3. Mucosal lesions BPDAI score accounts for ≥30% of total BPDAI activity score at randomisation
4. BP considered to be drug induced, in particular diagnosis of BP made within two months of starting a drug well known to induce BP
5. Treatment with BP-directed biologics including: a) Any cell-depleting agents including, but not limited to, rituximab within 12 months prior to baseline, b) Other biologics within five half-lives (if known) or 16 weeks prior to the baseline, whichever is longer, or c) Intravenous immunoglobulin within 16 weeks prior to the baseline.
6. Taking > 0.3 mg/kg/day OCS at screening
7. Treatment with systemic immunomodulators such as dapsone or doxycycline within four half-lives of the drugs prior to baseline Day 1
8. Treatment with immunosuppressants within the last two weeks prior to baseline
9. Treatment with an anti-complement therapy or with Zileuton within the last three months prior to baseline
10. OCS dose no more than 0.3mg/kg/day in the 7 days before screening visit
11. Taking super-potent topical corticosteroids and unable to discontinue them at or before the screening assessment
12. Active systemic or organ system bacterial or fungal infection or progressive severe infection
13. Known congenital immunodeficiency or a history of acquired immunodeficiency including a positive human immunodeficiency virus (HIV) test
14. Active infection with hepatitis B or C
15. Positive nasal throat swab for Neisseria species
16. Known hypersensitivity to nomacopan and any of its excipients
17. Receipt of live attenuated vaccines within 2 weeks of Day 1

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-05-06 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Achievement of Complete Disease Remission | weeks 16 - 24
  Proportion of patients in Complete Disease Remission

SECONDARY OUTCOMES:
Cumulative oral corticosteroid, OCS, during treatment | Randomization to 24 weeks
  Cumulative OCS used during treatment
Proportion of patients requiring rescue therapy | Randomization to 24 weeks
  Proportion of patients requiring rescue therapy during the 24 weeks of treatment
Achievement Partial Disease Remission | weeks 16 - 24
  Proportion of patients in Partial Disease Remission
Time to onset of Complete Disease Remission | week 6 to 24
  Time (weeks) to onset of Complete Disease Remission
Duration of Complete and Partial Disease Remission | week 6 to 24
  Duration (weeks) of Complete Disease Remission and Partial Disease Remission
Investigator Global Assessment (IGA) score | weeks 6 - 24
  Proportion of patients with Investigator Global Assessment (IGA) score of 0 or 1
Adverse Events | Day 1 to Week 28
  Frequency, type and relationship of AEs to treatment
Steroid-related AEs | Day 1 to Week 28
  Incidence of steroid-related AEs
Dermatology Life Quality Index (DLQI) | Randomisation to week 24
  Change from baseline in Dermatology Life Quality Index (DLQI)
Incidence of treatment-emergent anti-drug antibody (ADA) responses and titre and neutralising potential assessed in vitro at baseline and every 4 weeks | Day 1 to Week 28
  Incidence of treatment-emergent anti-drug antibody (ADA) responses and titre and neutralising potential assessed in vitro at baseline and then every 4 weeks

CONTACTS AND LOCATIONS:
Locations (12):
- United States (7):
  - Tulane University Health Sciences Center, Los Angeles, California
  - North Shore University Health System, Skokie, Illinois
  - Dawes Fretzin Clinical Research Group LLC, Indianapolis, Indiana
  - David Fivenson MD PLC, Ann Arbor, Michigan
  - Duke Dermatology, Durham, North Carolina
  - Wright State Physicians 725 University Blvd., Fairborn, Ohio
  - UMPC Department of Dermatology, Pittsburgh, Pennsylvania
- Germany (3):
  - MENSINGDERMA Research GmbH, Hamburg
  - Universitätsklinikum Schleswig-Holstein, Kiel
  - Universitäts Hautklinik, Tübingen
- University Medical Center Groningen, Groningen, Netherlands
- Cityclinic Przychodnia Lekarsko-Psychologiczna Matusiak Spółka Partnerska, Wroclaw, Poland

IPD SHARING:
Plan to Share IPD: No